CLINICAL TRIAL: NCT05304650
Title: A Usability Study of External Neuromodulation With iTEAR100 Generation 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olympic Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: clp 010
Record Dates: First submitted 2022-03-01; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- iTEAR100 Therapy (Other): Treatment Arm. Assessment of usability of generation 2 connected devices
  Interventions: Device: iTEAR100

INTERVENTIONS:
Device: iTEAR100 — Controlled Stimulation External Nasal Nerve to stimulate tear production

SUMMARY:
A Usability Study of External Neuromodulation With iTEAR100 Generation 2. A study which evaluates user ability to train and access the iTEAR100 device in a telehealth environment.

DETAILED DESCRIPTION:
A Usability Study of External Neuromodulation With iTEAR100 Generation 2. A study which evaluates user ability to train and access the iTEAR100 device in a telehealth environment. Subjects sign a consent form and are sent a device. After downloading a mobile app, they can access the device and download a prescription. At 7 days, an official telehealth visit evaluates their success in the set up and training. At 30 days, the trial ends, A usability survey and symptom evaluation survey are used to determine success.

ELIGIBILITY:
Inclusion Criteria: Able to sign English language consent form and over age 18 and reside in the U.S.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Usability | 30 days
  Subjects rate the device usability similar to daily mobile applications and home devices using a scale from -3 to +3 with 0 being same as every day devices such as bank application, restaurant application, etc.

SECONDARY OUTCOMES:
Symptom Scores | 30 days
  OSDI and SPEED standard symptom scores
Adverse Events | 30 days
  Skin Damage, Headache, Dizziness, Sneezing
Symptom Score | 30 Days
  SPEED standard symptom score

CONTACTS AND LOCATIONS:
Locations (1):
- Olympic Ophthalmics, Issaquah, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided